CLINICAL TRIAL: NCT02820506
Title: Sentinel Node Mapping With Robotic Assisted Near Infra-red Fluorescent Imaging in Women With Cervical and Endometrial Cancer
Brief Title: Sentinel Node Mapping in Women With Endometrial and Cervical Cancer
Acronym: SENTIREC II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Sara Sponholtz, MD, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SDUSF12015163 1 (198)1
Record Dates: First submitted 2016-06-23; First posted 2016-07-01 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Uterine Cervical Neoplasms; Uterine Neoplasms
Keywords: robotic surgery procedures; indocyanine green; sentinel lymph node mapping
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Intervention Model Description: Endometrial cancer, Diagnostic; Assessing the safety of the SLN mapping algorithm. Inclusion is defined by a power calculation: Assuming the true incidence of metastasis is 20% and the sensitivity of the SLN mapping algorithm is 96%. To obtain the conclusion that NPV is larger than 94% using a 95% two-sided exact Clopper-Pearson confidence interval, then 150 women with sentinel lymph node mapping, a FDG/PET-CT and Pelvic- and paraaortic lymph node dissection are needed.
  Cervical cancer: Study is diagnostic and primarily explorative.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High risk endometrial cancer (Other): Patients will receive sentinel node mapping, removal of PET-positive lymph nodes and finally conventional pelvic and paraaortic lymphadenectomy.
  Interventions: Procedure: SLN mapping and removal of PET-positive lymph nodes
- Cervical cancer tumor size 2-4 cm (Other): Patients will receive sentinel node mapping, followed by removal of PET-positive lymph nodes and finally conventional pelvic lymphadenectomy.
  Interventions: Procedure: SLN mapping and removal of PET-positive lymph nodes

INTERVENTIONS:
Procedure: SLN mapping and removal of PET-positive lymph nodes — Sentinel node mapping will be performed, followed by systematic removal og PET/CT positive lymph nodes

SUMMARY:
The aim of the study is to evaluate the feasibility of applying the SLN mapping technique in combination with FDG-PET/CT imaging in women with high-risk histology endometrial cancer and in patients with cervical cancer tumour size 2-4 cm.

ELIGIBILITY:
Inclusion Criteria:

* Study IIA: Patients with cervical cancer, FIGO IB1, tumor size 2-4 cm
* Study IIB: Patients with high risk endometrial cancer, presumed FIGO I, type 1 histology grade 3 Endometrioid adenocarcinoma or type 2 histology (serous-, clearcel-, carcinosarcoma or undifferentiated adenocarcinoma.

Exclusion Criteria:

* Prior PL
* Known allergy towards ICG and/or iodine (ICG contains 5% sodium iodine)
* Women included in other studies affecting outcome-measures of the present study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  Sensitivity of sentinel lymph node mapping compared to the sensitivity of sentinel lymph node mapping combined with removal of PET-positive lymph nodes
Negative predictive value | 2 years
  Negative predictive value of sentinel lymph node mapping algorithm, and a sentinel lymph node mapping algorithm including removal of PET-positive lymph nodes

SECONDARY OUTCOMES:
Specificity | 2 years
  Specificity of sentinel lymph node mapping compared to the combination of sentinel lymph node mapping and removal of PET-positive lymph nodes
Positive predictive value | 2 years
  Positive predictive value of sentinel lymph node mapping compared to the combination of sentinel lymph node mapping and removal of PET-positive lymph nodes
Prevalence of lymph node metastasis | 2 years
  Prevalence of lymph node metastasis in the pelvis and paraaortic area
Incidence of lymphedema | 3 years
  Using patient reported outcome measures
Severity of lymphedema | 3 years
  Using patient reported outcome measures
Quality of life rate | 3 years
  Using patient reported outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Pernille T Jensen, Professor, Principal Investigator — Aarhus University Hospital and Aarhus University, Denmark
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Bjornholt SM, Sponholtz SE, Markauskas A, Froding LP, Larsen CR, Fuglsang K, Schledermann D, Mogensen O, Jensen PT. Sentinel lymph node mapping for endometrial and cervical cancer in Denmark. Dan Med J. 2021 Mar 24;68(4):A11200886. PMID 33829991

DOCUMENTS (1):
  • Study Protocol (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT02820506/Prot_000.pdf